CLINICAL TRIAL: NCT05201651
Title: Effects of Creatine Supplementation on Motor Skill Acquisition and Related Neurophysiology
Brief Title: Creatine and Motor Skill Acquisition
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021-139
Record Dates: First submitted 2021-11-10; First posted 2022-01-21 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Young Healthy Adults (no Medical Condition/Disease)
Keywords: motor learning; transcranial magnetic stimulation; motor cortex; corticospinal excitability; creatine
MeSH Terms: conditions — Disease | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Participants assigned to receive creatine supplementation or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind. Individual without other involvement in study has study codes and prepares and distributes study kits containing creatine and placebo (similar appearance).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine (Experimental): Participants will orally consume creatine (20 grams in 4×5-gram servings for seven days), followed by 3-g/day during training days.
  Interventions: Dietary Supplement: Creatine Monohydrate
- Placebo (Placebo Comparator): Participants will orally consume maltodextrin placebo (20 grams in 4×5-gram servings for seven days), followed by 3-g/day during training days.
  Interventions: Dietary Supplement: Maltodextrin Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Participants will orally consume creatine (20 grams in 4×5-gram servings for seven days), followed by 3-g/day during training days. This 3-g/day dosage has been shown to maintain cellular creatine levels.
  Arms: Creatine
Dietary Supplement: Maltodextrin Placebo — Participants will orally consume maltodextrin placebo (20 grams in 4×5-gram servings for seven days), followed by 3-g/day during training days.
  Arms: Placebo

SUMMARY:
The investigators will conduct a double-blind, placebo-controlled, repeated measures study of the effects of oral creatine monohydrate supplementation on motor skill acquisition and neurophysiology in young healthy adults. After baseline testing, participants will be randomized to receive creatine supplementation or placebo for seven days. Participants will then complete three days of training on a motor skill task while consuming a maintenance dosage of creatine or placebo. TMS measures of neurophysiology will be assessed at baseline, and pre- and post-skill training on the first and third training days.

DETAILED DESCRIPTION:
Participants: Thirty-six young healthy adults between 18-39 years of age will participate in the study. Participants will follow an omnivore diet given differences in response to creatine supplementation among vegetarians.

Group allocation: Participants will be allocated to study groups (i.e., creatine, placebo) using blocked randomization that stratifies by sex (male, female).

Supplementation and diet: An individual blind to supplement and group allocation will prepare participant study kits. Each study kit will contain daily supplementation bags for the duration of the study, detailed instructions, and a compliance log. Creatine (Creapure® AlzChem Trostberg GmbH, Germany) and placebo (Globe Plus 10 DE Maltodextrin, Univar Canada) will be in powder form and be very similar in color, texture, and appearance. After baseline testing, participants will orally consume creatine or placebo (20 grams in 4×5-gram servings for seven days), followed by 3-g/day during training days. This 3-g/day dosage has been shown to maintain cellular creatine levels. Adherence with the supplementation protocol will be assessed by the compliance log. Possible adverse events to supplementation (i.e., minor gastrointestinal irritation) will be assessed using adverse event forms. Upon completion of the study, participants will be asked to guess whether creatine or placebo had been administered. Habitual dietary intake will be determined by 3-day food logs completed by participants prior to the study.

Motor skill task: Participants will perform an "intercept and release" task which uses a Microsoft Kinect sensor and open-source software to track 3-dimensional joint movement. Participants will be instructed to "save the world" through control of an on-screen cursor (i.e., spaceship) using movement of their dominant arm to intercept a moving object (an asteroid) as it emerges from the side of a computer screen. After interception of the object, participants will be required to accurately throw the object to hit a target (the sun). The task will progress through 10 stages of increasing difficulty (i.e., increasing object speed, decreasing target size) as skill performance improves. The stages of difficulty are designed to challenge participants, maintain engagement, and prevent plateaus in performance.

Participants will complete one block of 200 movements (i.e., 100 object interceptions, 100 object throws) at the easiest level of difficulty in the baseline testing session. After the initial 7-day creatine supplementation period, three training sessions will be completed on consecutive days. A training session will involve five blocks of 200 movements, for 1,000 skilled arm movements per session (~45 minutes), and a total of 3,000 training movements over the course of the study. A plot of object interception time (y-axis) by successful movement trial (x-axis) across the training period (i.e., days 1-3) will be generated for each participant and fit with an exponential curve. The curve fitting parameter that represents rate of skill acquisition will be extracted for each participant as the primary dependent variable.

Transcranial magnetic stimulation (TMS): Using neuronavigation software, TMS will be applied over the primary motor cortex to elicit motor evoked potentials (MEPs) in the extensor carpii radialis muscle of the dominant arm, a muscle involved in performance of the motor skill task. Using standard procedures, the investigators will collect a battery of TMS measures that provide indices of corticospinal excitability and gamma-aminobutyric acid and glutamate signaling at baseline, and pre- and post-skill training on the first and third days.

ELIGIBILITY:
Inclusion Criteria:

* omnivore diet

Exclusion Criteria:

* pre-existing liver abnormalities
* pre-existing kidney abnormalities
* pre-existing neuromuscular abnormalities
* contraindications to transcranial magnetic stimulation
* consumption of dietary supplements containing creatine within 30 days prior to the start of the study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of change in movement time | 3 days
  Both groups will perform a skill acquisition task that involves moving the dominant upper limb to direct a cursor towards moving targets presented on a computer screen. The task will be practiced over a period of three days. The time required to reach each moving target will be measured (i.e., movement time) with faster times indicating improved performance. The rate of improvement on the task over the three days will be determined.

SECONDARY OUTCOMES:
Single pulse motor evoked potential amplitude | Days 1 and 3 of training
  Amplitude of motor evoked potentials measured with electromyography and elicited by single-pulse transcranial magnetic stimulation. Provides a marker of corticospinal excitability.
Short-interval intracortical inhibition motor evoked potential amplitude | Days 1 and 3 of training
  Amplitude of motor evoked potentials measured with electromyography and elicited by transcranial magnetic stimulation using paired-pulse short interval intracortical inhibition paradigm.
Intracortical facilitation motor evoked potential amplitude | Days 1 and 3 of training
  Amplitude of motor evoked potentials measured with electromyography and elicited by transcranial magnetic stimulation using paired-pulse intracortical facilitation paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron S Mang, PhD, Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
Will not share individual participant data.